CLINICAL TRIAL: NCT03365310
Title: Clinical Evaluation of Turmeric and Tulsi Polyherbal Formulation in the Management of Frailty in Elderly Population: An Open Label Randomized Controlled Trial
Brief Title: Management of Frailty in Older Adults With Turmeric and Tulsi Supplements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Composite Interceptive Med Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OI-007-2017
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Frail Elderly Syndrome
MeSH Terms: interventions — Diarylheptanoids; Milk; holy basil leaf extract; Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel follow up of two treatment groups randomly allocated through a central randomization process
Masking Description: open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive turmeric and tulsi capsule with milk(100 ml) along with standard of care treatment as determined by research physician...Each participants has to take two capsules of turmeric formula and tulsi twice daily for the study period of 3 months
  Interventions: Drug: C. longa, curcuminoids , Z. officianale, O. sanctum along with 200 ml of Milk; Other: Standard of Care
- Standard Care Group (Active Comparator): Participants will only receive the standard of care treatment as determined by research physician
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: C. longa, curcuminoids , Z. officianale, O. sanctum along with 200 ml of Milk — Polyherbal formulation along with standard of care
  Other Names: Turmeric formula and Tulsi capsule and Milk
  Arms: Intervention Group
Other: Standard of Care — Usual standard of care for consist of exercise, caloric and protein support, vitamin D, reduction of polypharmacy along with medical management of health condition, assessment of care needs and provision of care. These will be determined on case by case basis by research clinician.

SUMMARY:
The aim of this study is to determine the efficacy of turmeric and tulsi polyherbal formulation in the management of frailty in the elderly population.

DETAILED DESCRIPTION:
Frailty is a wasting syndrome of old age that leaves a person vulnerable to falls, functional decline, morbidity and mortality. Reducing the severity of frailty will provide large benefits for individuals, their families and for the society. It is assumed that early intervention with frail people will improve quality of life and reduce the costs of care. This trial is testing the frailty intervention with herbal medicine. If this frailty intervention is shown to be effective, there are major potential benefits to the frail older population generally in terms of decreased disability. The interventions being examined are readily transferable to routine clinical practice and can potentially be applied routinely in aged care services.

ELIGIBILITY:
Inclusion Criteria:

* Subjects above the age of 65 years, providing written informed consent.
* Meeting three or more Cardiovascular health study frailty criteria
* Mild or no cognitive impairment (defined as a Mini-Mental State Examination score >23),
* Able to walk without personal assistance and no other physical limitations that can limit participation and adherence, particularly to exercise intervention program

Exclusion Criteria:

People will be ineligible to participate in the trial if they:

* Live in a residential aged care facility
* Severe audio-visual impairment
* Progressive, degenerative neurologic disease like Parkinsonism, fits/ epilepsy, etc.
* Rapidly progressive or terminal illness under palliative care with life expectancy less than 12 months
* History of alcohol abuse or any other substance abuse
* Severely affect muscle/joint dysfunction resulting in disability
* Hospital admission in the past 3 months
* Regular physical training or physiotherapy or current participation in a vigorous exercise or weight-training program more than once per week
* Undergoing therapeutic diet incompatible with nutritional supplementation
* In the opinion of research clinician, the intervention is deemed to be potentially hazardous for the subject, such as serious cardiac and pulmonary disease.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Frailty Score | 3 months
  To assess a change in frailty score from baseline in 3 months between two groups

SECONDARY OUTCOMES:
C reactive protein | 3 months
  Change in C-reactive Protein (CRP) from baseline
Frequency of falls | 3 months
  defined as an event resulting in a person coming to rest unintentionally on the ground or other lower level; near-falls would not be included
Health service utilization | 3 months
  frequencies of doctor visits, emergency room visit, hospitalization, nursing home admission
Mortality | 3 months
  Death of study participant during study period

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjaya Chauhan, Principal Investigator — Composite Interceptive Med Science; Dr. Alben Sigamani, Principal Investigator — Narayana Hrudayalaya Hospital
Locations (1):
- Mazumdar Shaw Medical Centre, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided